Protocol Number: 20200392

Product: AMG 176

Date: 10 May 2024 

#### **Statistical Analysis Plan**

| Protocol Title: | A Phase 1 Study of AMG 176 as Monotherapy and in Combination with Azacitidine in Higher-Risk Myelodysplastic Syndrome and Chronic Myelomonocytic Leukemia. | |
|---|---|---|
| Short Protocol Title: | Phase 1 Study of AMG 176 w<br>Subjects with MDS/CMML | ith Azacitidine in |
| Protocol Number: | 20200392 | |
| NCT Number: | Not available at the time of an | nendment |
| Authors: | | |
| Sponsor: | Amgen, Inc. | |
| | One Amgen Center Drive | |
| | Thousand Oaks, CA 91320 | |
| SAP Date: | Document Version [ | <u>Date</u> |
| | Amendment 1 (v2.0) | 10 May 2024 |

| Version Number | Date<br>(DDMMMYYYY) | Summary of Changes, including rationale for changes |
|---|---|---|
| Original (v1.0) | 20OCT2021 | Original Version |
| Amendment 1 (v2.0) | 10MAY2024 | <ul> <li>CMML is added along with R/R MDS in the secondary objectives.</li> <li>Secondary endpoint 'Evaluate the pharmacokinetics (PK) of the AMG 176 when administered as monotherapy' is added.</li> <li>Overall response according to Uniform Response Criteria is now changed to overall response according to International Working Group (2006) -MDS/MPN Response criteria throughout the SAP except for objectives and endpoints.</li> </ul> |



Protocol Number: 20200392

Date: 10 May 2024 

| • | The description for Part 1 changed |
|---|-------------------------------------|
| | from 'Dose Escalation/ |
| | Determination of Maximum |
| | Tolerated Combination Dose |
| | (MTCD) and Recommended |
| | Phase 2 Dose (RP2D)' to 'Dose |
| | Escalation/Determination of Optimal |
| | Biological Dose (OBD) and |
| | Minimum Safe and Biologically |
| | Effective Dose (MSBED) |

- Two dose levels in part 1 changed to three dose levels.
- The text of MTDC/RP2D definition is now replaced with 'The DLRT may change the dose/dosing scheduled based on emerging data. The OBD/MSBED is defined as the minimum safe and biologically effective combination dose with a probability of DLT lower than or close to a targeted toxicity probability of 0.2'
- In Part 2 the enrollment in newly diagnosed subjects is changed as 'subjects will not be enrolled into this cohort until all previous cohorts have been completed and the data reviewed by the FDA. Toxicity will be monitored for each cohort using a Bayesian approach proposed by Thall, Simon, and Estey (1995).'
- Prior distribution parameters are changed to beta (1,1) whereas initially it was beta (0.50, 1.50).
- The posterior probability that the incidence is greater than 30% is > 90% is changed to '20% is greater than 80%.
- The sample size changed from 110 subjects to 120 subjects and number of subjects in part 1 changed from 50 to 60
- BOR definition is updated as BOR is defined as the first response category achieved as responders and non-responders. Responders will include CR or PR, whereas



Protocol Number: 20200392

Date: 10 May 2024 

| non-responders will include SD,<br>PD, NE or NA. |
|---|
| <ul> <li>Section 10- changes from protocol specified analysis is updated.</li> </ul> |
| <ul> <li>Section 9.1- Updated the general considerations.</li> </ul> |
| <ul> <li>Section 9.5.2- Updated to<br/>include listings for<br/>responder/non-responder.</li> </ul> |



Protocol Number: 20200392

Date: 10 May 2024

#### **Table of Contents**

| Tab | le of C | ontents | 4 |
|---|---|---|---|
| 1. | Introd | duction | 11 |
| 2. | Obje | ctives, Endpoints/Estimands and Hypotheses | 11 |
| | 2.1 | Objectives and Endpoints/Estimands | |
| | 2.2 | Hypotheses and/or Estimations | |
| 3. | Study | / Overview | 12 |
| | 3.1 | Study Design | |
| | 3.2 | Sample Size | |
| | 3.3 | Adaptive Design | |
| 4. | Cova | riates and Subgroups | 15 |
| | 4.1 | Planned Covariates | |
| | 4.2 | Subgroups | |
| 5. | Defin | itions | 15 |
| 6. | | vsis Sets | |
| 0. | 6.1 | Full Analysis Set. | |
| | 6.2 | DLT Evaluable Analysis Set | |
| | 6.3 | Pharmacokinetic/Pharmacodynamic Analyses Set(s) | |
| 7. | | ned Analyses | |
| 1. | 7.1 | Interim Analysis and Early Stopping Guidelines | |
| | 7.1 | Primary Analysis | |
| | 7.2 | Final Analysis | |
| | | • | |
| 8. | | Screening and Acceptance | |
| | 8.1 | General Principles | |
| | 8.2 | Data Handling and Electronic Transfer of Data | |
| | 8.3 | Handling of Missing and Incomplete Data | |
| | 8.4 | Detection of Bias | |
| | 8.5 | Outliers | |
| | 8.6<br>8.7 | Distributional Characteristics | |
| | | • | |
| 9. | | stical Methods of Analysis | |
| | 9.1 | General Considerations. | |
| | 9.2 | Subject Accountability | |
| | 9.3 | Important Protocol Deviations | |
| | 9.4 | Demographic and Baseline Characteristics | |
| | 9.5 | Efficacy Analyses | |
| | | 9.5.1 Analyses of Primary Efficacy Endpoint(s)/Estimand(s) | 21 |



Protocol Number: 20200392

| Date: | 10 May 2024 | Page 5 of 3 |
|-------|-------------|-------------|

| | | 9.5.2 | Analyses of Secondary Efficacy Endpoint(s)/Estimand(s) | 21 |
|---|---|---|---|---|
| | | 9.5.3 | Analyses of Exploratory Efficacy Endpoint(s) | |
| | 9.6 | Safety A | Analyses | |
| | | 9.6.1 | Analyses of Primary Safety Endpoint(s) | 21 |
| | | 9.6.2 | Adverse Events | 21 |
| | | 9.6.3 | Laboratory Test Results | 21 |
| | | 9.6.4 | Vital Signs | 22 |
| | | 9.6.5 | Physical Measurements | 22 |
| | | 9.6.6 | Electrocardiogram | 22 |
| | | 9.6.7 | Antibody Formation | 22 |
| | | 9.6.8 | Exposure to Investigational Product | 22 |
| | | 9.6.9 | Exposure to Non-investigational Product(s)/Auxiliary Medicinal Product(s) | 22 |
| | | 9.6.10 | Exposure to Concomitant Medication | 22 |
| | 9.7 | Other A | nalyses | 22 |
| | | 9.7.2 | Analyses of Pharmacokinetic or Pharmacokinetic/Pharmacodynamic Endpoints | 22 |
| | | 9.7.3 | Analyses of Clinical Outcome Assessments | 22 |
| | | 9.7.4 | Analyses of Health Economic Endpoints | 23 |
| 10. | Chan | ges From | Protocol-specified Analyses | 23 |
| 11. | Litera | ature Citati | ons / References | 24 |
| 12. | Priori | tization of | Analyses | 26 |
| 13. | Data | Not Cover | ed by This Plan | 26 |
| 14. | Appe | ndices | | 27 |
| | Appe | ndix A. C | ode Fragments | 27 |
| | Appe | ndix B. M | odified Toxicity Probability Interval Design | 28 |
| | | | ast Known Alive Date | |
| | Appe | ndix D. H | andling of Dates, Incomplete Dates and Missing Dates | 31 |
| | Appe | ndix E. MI | OS Diagnostic and Response Criteria | 33 |



Protocol Number: 20200392

Date: 10 May 2024 

#### **List of Abbreviations**

| Abbreviation | Explanation |
|---|---|
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ALT | alanine aminotransferase |
| AML | acute myeloid leukemia |
| ANC | absolute neutrophil count |
| AST | aspartate aminotransferase |
| ASTX727 | Cedazuridine |
| AUC | area under the curve |
| BAK | pro-apoptotic effector proteins BCL2 homologous antagonist/killer |
| BAX | pro-apoptotic effector proteins BCL2-associated X |
| BCL2 | B-cell lymphoma/leukemia 2 |
| BCRP | breast cancer resistance protein |
| ВН3 | pro-apoptotic BCL2 homology 3 |
| BIM | BCL2-interacting mediator of cell death |
| BUN | blood urea nitrogen |
| CC-486 | Azacitidine |
| CFR | U.S. Code of Federal Regulations |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK-MB | creatine kinase-muscle/brain |
| CL | Clearance |
| C <sub>max</sub> | maximum concentration |
| CMML/CMMoL | chronic myelomonocytic leukemia |
| COVID-19 | Coronavirus Disease 2019 |
| CR | complete remission |
| CrCl | creatinine clearance |
| CRF | case report form |
| CRi | incomplete count recovery |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CYP | cytochrome P450 |
| DDI | drug-drug interaction |
| DILI | drug induced liver injury |
| DLRM | dose level review meeting |
| DLRT | dose level review team |



Protocol Number: 20200392

Date: 10 May 2024 

DLT dose limiting toxicity
DOR duration of response
DR durable response
ECG Electrocardiogram
Echo Echocardiogram

ECOG PS Eastern Cooperative Oncology Group Performance Status

eCRF electronic case report form

EDC electronic data capture

EFS event-free survival

EOS end of study

EOT end of treatment

FAB French – American – British subtypes

FAS full analysis set

FDA Food and Drug Administration

FIH first in human

FSH follicle-stimulating hormone

GCP Good Clinical Practice

G-CSF granulocyte-colony stimulating factor

GLP good laboratory practices
GSO Global Safety Officer
HALs Houston Area Locations
HbcAb hepatitis B core antibody
HbsAb hepatitis B surface antibody
HbsAg hepatitis B surface antigen
HCVAb hepatitis C virus antibody

hERG human ether-à-go-go-related gene

Hgb Hemoglobin

HI hematologic improvement

HIPAA Health Insurance Portability and Accountability Act

HIV human immunodeficiency virus

HMA hypomethylating agent

HNSTD highest-non-severely-toxic dose

HR higher-risk

HSCT hematopoietic stem cell transplant

IB Investigator's Brochure

IC50 half-maximal inhibitory concentration



Protocol Number: 20200392

Date: 10 May 2024 

ICF informed consent form

ICH International Council for Harmonisation

ICJME International Committee of Medical Journal Editors

IEC Independent Ethics Committee

IND Investigational New Drug
INR international normalized ratio

IPSS International Prognostic Scoring System

IPSS-R Revised IPSS

IRB Institutional Review Board

IRT interactive response technology
ISS International Staging System

ITT intent-to-treat

IUD intrauterine device

IUS intrauterine hormonal-releasing system

IV Intravenous

Ki mean inhibitory constant

KM Kaplan-Meier

LDH lactate dehydrogenase

LVEF left ventricular ejection fraction
MAD maximum administered dose

MCL1 Myeloid Leukemia Cell 1

mCR marrow/morphologic complete remission

MDS myelodysplastic syndrome

MDSCs Myeloid Derived Suppressor Cells

MM Multiple Myeloma

MOA mechanism of action

MOLM acute monocytic leukemia (AML-M5a) cell lines

MOMP mitochondrial outer membrane permeabilization

MPN myeloproliferative neoplasm

MPN-SAF MPN Symptoms Assessment Form

MRD minimum residual disease

MRI magnetic resonance imaging

MSBED minimum safe and biologically effective dose

mTPI modified Toxicity Probability Interval

MUGA scan Multigated Acquisition scan
NCI National Cancer Institute

Protocol Number: 20200392

Date: 10 May 2024 

NCT National Clinical Trials

NE Not evaluable

NK cells natural killer cells

NT-pro BNP N-terminal prohormone of brain natriuretic peptide

NYHA New York Heart Association

OATP organic anion polypeptide transporters

OBD optimal biological dose
ORR overall response rate

OS overall survival

PBMC peripheral blood mononuclear cell

PCR polymerase chain reaction

PD progressive disease

PFS progression free survival

PI principal investigator
PK Pharmacokinetics

PLT Platelets

PR partial remission

PUMA p53-upregulated modulator of apoptosis

Q2W every 2 weeks

QD2 once daily for 2 consecutive days

QRS QRS interval is the interval between the Q wave and the S wave

in the heart's electrical cycle as measured by ECG; represents

the time it takes for the depolarization of the ventricles

QTc corrected QT interval

QTcF QT interval with Fridericia's correction

QW once weekly

R/R relapsed or refractory
RA refractory anemia

RAEB refractory anemia with excess blasts

RAEB-T refractory anemia with excess blasts in transformation

RARS refractory anemia with ringed sideroblasts

RBC red blood cell

SAP statistical analysis plan

SC Subcutaneous
SD stable disease

siRNA small interfering RNA



Protocol Number: 20200392

Date: 10 May 2024 

SOC standard of care

STD severely-toxic dose

t<sub>1/2</sub> half-life

TBL total bilirubin

TI transfusion independence

TLS tumor lysis syndrome
TSS Total Symptom Score
TTNT time to next treatment
ULN upper limit of normal
UPM Unit Probability Mass
URL Upper Reference Limit

USPI United States Prescribing Information

Ven Venetoclax

WBC white blood cells

WHO World Health Organization

WHODRUG World Health Organization Drug

Protocol Number: 20200392

Date: 10 May 2024 

#### 1. Introduction

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within the **protocol superseding amendment 3** for study 20200392, AMG 176 dated **28 April 2022**. The scope of this plan includes the final analysis that is planned and will be executed by the Amgen Global Biostatistical Science department unless otherwise specified.

#### 2. Objectives, Endpoints/Estimands and Hypotheses

#### 2.1 Objectives and Endpoints/Estimands

| Objectives | Endpoints |
|---|---|
| Primary | |
| Part 1A – QW Monotherapy (Dose Exploration) Evaluate the safety and tolerability of AMG 176 once weekly (QW) monotherapy in subjects with R/R higher risk myelodysplastic | Incidence of dose limiting toxicities<br>(DLTs), treatment-related,<br>treatment-emergent adverse events<br>and clinically significant changes in |
| syndrome (HR-MDS) | vital signs, electrocardiogram (ECGs),<br>and clinical laboratory tests |
| Part 1B – QW Combination Therapy (Dose | · |
| <ul> <li>Evaluate the safety and tolerability of<br/>AMG 176 in combination with<br/>azacitidine in subjects with R/R<br/>HR-MDS and determine the Optimal<br/>Biological Dose (OBD) and Minimum<br/>Safe and Biologically Effective Dose<br/>(MSBED) of AMG 176 in combination<br/>with azacitidine</li> </ul> | Incidence of DLTs, treatment-related,<br>treatment-emergent adverse events<br>and clinically significant changes in<br>vital signs, ECGs, and clinical<br>laboratory tests |
| Part 2 – QW Combination Therapy (Dose Expan | nsion) |
| Evaluate the preliminary efficacy of AMG 176 in combination with azacitidine in subjects with R/R HR-MDS/CMML in: LIMA Failure, Venetagley New York | Overall response rate (ORR),<br>according to the Uniform Response<br>Criteria for Myelodysplastic/<br>Myeloproliferative Neoplasms<br>(MDS/MPN), including: |
| HMA Failure, Venetoclax-Naïve HMA Failure, Venetoclax Expanded. | Complete Remission (CR) |
| <ul> <li>HMA Failure, Venetoclax-Exposed</li> <li>To assess the preliminary efficacy of<br/>AMG 176 in combination with</li> </ul> | Partial Remission (PR) Marrow CR |
| azacitidine in subjects with Newly<br>Diagnosed MDS/CMML | Cytogenic response |

#### **Secondary**

Part 1A – QW Monotherapy (Dose Exploration)

Protocol Number: 20200392

Date: 10 May 2024 

| Evaluate preliminary efficacy of<br>AMG 176 QW when given as<br>monotherapy in R/R MDS/CMML | Overall response according to the<br>Uniform Response Criteria for<br>MDS/MPN, Event-Free Survival<br>(EFS), time to response, and Duration<br>of Response (DOR) |
|---|---|
| Evaluate the pharmacokinetics<br>(PK) of AMG 176 when<br>administered as monotherapy | PK parameters for AMG 176 including, but not limited to, maximum observed concentration (C <sub>max</sub> ), area under the concentration-time curve (AUC), clearance (CL), and half-life (t <sub>1/2</sub> ) |
| Part 1B – QW Combination Therapy (Dose Exp | loration) |
| Evaluate preliminary efficacy of<br>AMG 176 QW in combination with<br>azacitidine in R/R MDS/CMML | Overall response according to the<br>Uniform Response Criteria for<br>MDS/MPN, EFS, time to response,<br>and DOR |
| Evaluate the PK of AMG 176 and<br>azacitidine when administered in<br>combination | PK parameters for AMG 176 and azacitidine including, but not limited to, C <sub>max</sub> , AUC, CL, and t <sub>1/2</sub> |
| Part 2 – QW Combination Therapy (Dose E | xpansion) |
| Evaluate the preliminary efficacy of<br>AMG 176 in combination with<br>azacitidine in subjects with<br>R/R HR-MDS/CMML in: | Time to transformation to Acute Myeloid Leukemia (AML) Duration of Response (DOR) |
| <ul> <li>HMA Failure, Venetoclax-Naïve</li> <li>HMA Failure, Venetoclax-Exposed</li> <li>To assess the preliminary efficacy of AMG 176 in combination with azacitidine in subjects with Newly Diagnosed MDS/CMML</li> </ul> | <ul> <li>Overall Survival (OS)</li> <li>Time to Next MDS Treatment (TTNT)</li> <li>EFS</li> </ul> |
| Evaluate the PK of AMG 176 and azacitidine when administered in combination | PK parameters for AMG 176 and azacitidine including, but not limited to, C <sub>max</sub> , AUC, CL, and t <sub>1/2</sub> |

#### 2.2 Hypotheses and/or Estimations

The clinical hypothesis is that at least 1 dose level of AMG 176 administered in combination with azacitidine will achieve acceptable safety and tolerability in subjects with HR-MDS. No formal statistical hypothesis will be tested.

#### 3. Study Overview

#### 3.1 Study Design

This study is a phase 1 clinical trial designed to assess the safety, tolerability, and efficacy of AMG 176 as monotherapy and in combination with the 7-day regimen of



Protocol Number: 20200392

Date: 10 May 2024 

azacitidine for the treatment of HR-MDS/CMML. Subjects will be treated with Intravenous (IV) AMG 176 and IV or Subcutaneous (SC) azacitidine. The study consists of two parts.

### Part 1 – Dose Escalation/Determination of Optimal Biological Dose (OBD) and Minimum Safe and Biologically Effective Dose (MSBED)

In Part 1, the modified Toxicity Probability Interval (mTPI) design will be applied for dose escalation.

Three dose levels of AMG 176 monotherapy will first be tested in Part 1A, and after the OBD or MSBED is found, three dose levels of AMG 176 in combination with azacitidine will be tested in Part 1B.

Each dose cohort will initially enroll 3 to 4 subjects and up to 10 subjects per cohort may be enrolled. After reviewing all available safety data, dose level recommendations (eg, escalation, de-escalation) will be made by the Dose Level Review Team (DLRT) using an mTPI model (Ji et al, 2010) based on all subjects that have been enrolled at the current dose. The DLRT may change the dose/dosing scheduled based on emerging data. The OBD/MSBED is defined as the minimum safe and biologically effective combination dose with a probability of DLT lower than or close to a targeted toxicity probability of 0.2.

Dose escalation is considered complete if one of the following rules is met:

- 1. The highest planned dose level is evaluated, OBD has not been defined, and no DLTs occur at any dose level. In this case, the Maximum Administered Dose (MAD) may be used for Part 2.
- 2. An OBD is identified.

Guidelines for dose level decisions can be found in Table 3-1. Details regarding the mTPI model are described in Appendix B.

Table 3-1. Guidelines for Dose Level Decisions in Part 1

| | Number of DLTs | | |
|---|---|---|---|
| No. of DLT-evaluable <sup>a</sup> subjects treated at current dose | Escalate | Stay at current dose | De-escalate <sup>b</sup> |
| 3 | 0 | 1 | ≥ 2 |
| 6 | 0-1 | - | ≥ 2 |
| 9 | 0-1 | 2 | ≥ 3 |



Protocol Number: 20200392

Date: 10 May 2024 

| | Number of DLTs | | |
|---|---|---|---|
| No. of DLT-evaluable <sup>a</sup> subjects treated at current dose | Escalate | Stay at current dose | De-escalate <sup>b</sup> |
| 10° | 0-1 | 2-3 | ≥ 4 |

DLT = dose limiting toxicity.

#### Part 2 – Dose Expansion (Not Applicable, did not enroll)

Upon completion of Part 1 of the study, the dose expansion phase will begin at the **OBD/MSBED** and drug administration schedule with the intention of confirming the safety and tolerability and determining the efficacy of AMG 176 in combination with azacitidine in not only R/R HR- MDS/CMML, but also in frontline HR-MDS/CMML. An additional 60 subjects will be enrolled in Part 2 of the study as follows:

- HMA Failure Cohort: stratified by venetoclax exposure history
  - HMA Failure, venetoclax-Naïve (n = 20)
  - HMA Failure, venetoclax-Exposed (n = 20)
- Newly Diagnosed (n = 20) subjects will not be enrolled into this cohort until all previous cohorts have been completed and the data reviewed by the FDA.
   Toxicity will be monitored for each cohort using a Bayesian approach proposed by Thall, Simon, and Estey (1995).

The incidence of grade 3 or higher treatment-related non-hematological adverse events will be evaluated once every 5 subjects have had the chance to receive at least 1 cycle of treatment at the determined dose level for Part 2. Assuming a prior distribution of beta (1, 1), if the posterior probability that the incidence is greater than 20% is > 80% at these interim analyses, the study will stop early. The purpose of the safety interim analyses is to assess if the threshold for early termination has been reached. The stopping rules and operating characteristics are described in Protocol Table 3-2 and Table 3-3.

Table 3-2. Stopping Boundary for Each Cohort in Part 2

| Number of subjects | Stop study if observing this number of subjects with grade 3 or higher treatment-related non-hematological adverse event |
|---|---|
| 5 ~ 6 | ≥ 2 |



<sup>&</sup>lt;sup>a</sup> A subject is considered DLT-evaluable if he/she experienced a DLT during the DLT evaluation period; or if he/she received 75% of the planned doses of AMG 176 and 100% of the planned doses of azacitidine and completed the DLT evaluation period.

<sup>&</sup>lt;sup>b</sup> De-escalate guideline applies only when current dose level and enrollment is allowed to a lower dose level.

<sup>&</sup>lt;sup>c</sup> The maximum number of evaluable subjects at one dose level is 10.

Protocol Number: 20200392

Date: 10 May 2024 

| 7 ~ 10 | ≥ 3 |
|---------|-----------|
| 11 ~ 14 | ≥ 4 |
| 15 ~ 19 | ≥ 5 |
| 20 | Completes |

Table 3-3. Operating Characteristics in Part 2

| True grade 3 or higher treatment-related non-hematological adverse event rate | Probability of early stopping |
|---|---|
| 0.10 | 15% |
| 0.15 | 32% |
| 0.20 | 51% |
| 0.25 | 69% |
| 0.30 | 82% |

#### 3.2 Sample Size

It is anticipated that up to 120 subjects will be enrolled in the study, with up to 60 subjects in Part 1 and 60 subjects in Part 2.

For each part, the sample size is based on practical considerations **and it is consistent** with conventional oncology studies with the objective to identify the OBD/MSBED.

#### 3.3 Adaptive Design

NA

#### 4. Covariates and Subgroups

#### 4.1 Planned Covariates

There are no planned covariates in this study.

#### 4.2 Subgroups

There are no planned subgroups in this study.

#### 5. Definitions

#### **Age at Enrollment:**

Age at Enrollment: Subject age at enrollment will be collected in [years] in the clinical database



Protocol Number: 20200392

Date: 10 May 2024 

#### Baseline:

Unless otherwise specified, baseline will be defined as the last assessment with nonmissing value before the first dose of investigational product (AMG 176).

#### **Baseline and Post-Baseline ECG Values in Triplicate:**

The baseline ECG is defined as the mean of all pre-dose assessments, the mean of values in a triplicate should be calculated before taking the mean of the triplicate averages.

For all post-baseline ECG, the mean value for measurements taken at the same assessment will be calculated and used in the analysis.

When an ECG is missing within a triplicate, all available data will be averaged for that time point.

#### **Bazett-corrected QT Interval (QTcB):**

The Bazett correction will be calculated from the investigator reported QT (msec) and RR interval (msec): QTcB=QT/(RR/1000)<sup>1/2</sup>

#### Best Overall Response (BOR):

BOR for a subject is the best observed post-baseline disease response based on investigator assessment.

BOR is defined as the first response category achieved as responders and non-responders. Responders will include CR or PR, whereas non-responders will include SD, PD, NE or NA.

Response criteria to be used for MDS/**MPN** are International Working Group (**IWG**)-**MDS** Response Criteria (2006).

#### Change From Baseline:

Change from baseline is the arithmetic difference between post-baseline and baseline.

#### **Duration of Treatment:**

Date of last administration of investigational product – Study Day 1 + 1



Protocol Number: 20200392

Date: 10 May 2024 

#### **DLT Observation Period:**

The DLT observation period is defined as day 1 through day 28 after the administration of the first dose of AMG 176.

#### Fridericia-corrected QT Interval (QTcF):

The Fridericia correction will be calculated from the investigator reported QT (msec) and RR interval (msec): QTcF=QT/(RR/1000)1/3.

#### <u>Investigational Product (IP):</u>

IP is used in reference to AMG 176.

#### Last known alive date:

Last known alive date is described in Appendix C.

#### Study Day:

Post study day 1: study day = (date – date of Study Day 1) + 1

Pre study day 1: study day = (date – date of Study Day 1)

#### Study Day 1:

Study day 1 is defined as the first day of administration of the investigational product after enrollment. The day prior to Study Day 1 is considered Day -1.

#### **Transfusion independence:**

Transfusion independence is defined as no transfusion for at least 8 consecutive weeks (56 days).

#### <u>Treatment-Emergent Adverse Event (TEAE):</u>

A treatment-emergent adverse event is any adverse event starting on or after the first dose of investigational product, as determined by "Did event start before first dose of investigational product" equal to "No" or missing on the Events eCRF, and up to and including 30 days after the last dose of investigational product excluding events reported after end of study date.

#### <u>Treatment-related Treatment-emergent Adverse Event (TRAE):</u>

A TRAE is any TEAE whose causal relationship is marked as "Related" on the eCRF.



Protocol Number: 20200392

Date: 10 May 2024 

Event with missing relationship will be assumed to be treatment-related.

#### 6. Analysis Sets

#### 6.1 Full Analysis Set

The FAS is defined as all subjects who are enrolled and receive at least 1 dose of AMG 176.

#### 6.2 DLT Evaluable Analysis Set

Subjects are considered DLT-evaluable if they experience a DLT during the DLT evaluation period, or if they complete the DLT evaluation period and receive at least 75% of the planned doses of AMG 176 and 100% of the planned dose of azacitidine.

#### 6.3 Pharmacokinetic/Pharmacodynamic Analyses Set(s)

The PK Analysis Set defined as all subjects who have received at least 1 dose of the investigational product and have at least 1 PK sample collected. These subjects will be evaluated for PK analysis unless the number of data points required for analysis is not enough, or significant protocol deviations have affected the data, or if key dosing or sampling information is missing.

#### 7. Planned Analyses

#### 7.1 Interim Analysis and Early Stopping Guidelines

As the decision was made to terminate the study early, no formal interim analysis will be performed for this study.

#### 7.2 Primary Analysis

No formal primary analysis will be performed due to early close out of the study.

#### 7.3 Final Analysis

A final analysis is planned after all available subjects have had the opportunity to complete the last study visit.

#### 8. Data Screening and Acceptance

#### 8.1 General Principles

The objective of the data screening is to assess the quantity, quality, and statistical characteristics of the data relative to the requirements of the planned analyses.



Protocol Number: 20200392

Date: 10 May 2024 

#### 8.2 Data Handling and Electronic Transfer of Data

The Amgen Global Study Operations-Data Management (GSO-DM) department will receive and store all data to be used in the planned analyses. This study will use the RAVE database.

#### 8.3 Handling of Missing and Incomplete Data

The following imputation for missing or incomplete data will be performed if required: Incomplete adverse event and concomitant medication dates missing data will be imputed as described in Appendix D.

Non-pharmacokinetic measurements ( ) that are above or below the quantification limits will be considered equal to the upper or lower limit of quantification for all analyses unless specified otherwise.

#### 8.4 Detection of Bias

Lack of protocol compliance and the potential for biased statistical analyses will be examined by assessing the incidence of important protocol deviations in each cohort.

The clinical study team will identify and document the criteria for important protocol deviations.

#### 8.5 Outliers

Outlier data will not be excluded unless scientifically justified.

PK concentration data will be evaluated for outliers by visual inspection and decisions to re-assay individual samples will be made in accordance with standard Pharmacokinetics and Drug Metabolism (PKDM) practices.

#### 8.6 Distributional Characteristics

Where appropriate, the assumptions underlying the proposed statistical methodologies will be assessed. If required data transformations or alternative non-parametric methods of analyses will be utilized.

#### 8.7 Validation of Statistical Analyses

Datasets, tables, figures, and listings will be produced and validated in accordance with SOP-430399. Standard macros will be used when available.



Protocol Number: 20200392

Date: 10 May 2024 

The production environment for statistical analyses consists of Amgen-supported versions of statistical analysis software; for example, the SAS System version 9.2 or later.

#### 9. Statistical Methods of Analysis

#### 9.1 General Considerations

Descriptive statistics on required continuous data like Troponin I and Troponin T will include means, medians, standard deviations, first and third quartiles and ranges.

When data are summarized by time, the values recorded against the scheduled time points listed in the protocol will be used. When assessing minimum/maximum increases or decreases over the study, all assessments, including unscheduled assessments will be used.

No formal statistical analysis will be performed for the study and listings will be provided.

#### 9.2 Subject Accountability

No summary of subject accountability will be required to provided.

#### 9.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined by the study team before the first subject's initial visit and updated during the IPD reviews throughout the study prior to database lock. These definitions of IPD categories, subcategory codes, and descriptions will be used during the course of the study. Eligibility deviations are defined in the protocol.

No listing of IPDs and eligibility deviations will be provided

#### 9.4 Demographic and Baseline Characteristics

Demographic and baseline characteristic will be listed.



Protocol Number: 20200392

Date: 10 May 2024 

#### 9.5 Efficacy Analyses

#### 9.5.1 Analyses of Primary Efficacy Endpoint(s)/Estimand(s)

No formal statistical analyses will be performed for primary efficacy endpoints due to early termination of the study which resulted in insufficient number of subjects.

## 9.5.2 Analyses of Secondary Efficacy Endpoint(s)/Estimand(s) The listing of responder/non-responder will be provided for Part 1A- QW Monotherapy (Dose Exploration) subjects.

#### 9.5.3 Analyses of Exploratory Efficacy Endpoint(s)

NA

#### 9.6 Safety Analyses

#### 9.6.1 Analyses of Primary Safety Endpoint(s)

No summary analysis tables will be provided for the safety endpoints. More details are mentioned in sections from 9.6.2 to 9.6.10

#### 9.6.2 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) version 26.1 or later will be used to code all events categorized as adverse events to a system organ class and a preferred term.

Subject listing of all treatment-emergent adverse events, serious adverse events, adverse events leading to discontinuation of investigational product, treatment related adverse events, DLTs and fatal adverse events will be provided.

Subject listing of Troponin increased adverse events serious adverse events, adverse events leading to discontinuation of investigational product, treatment related adverse events, and fatal adverse events will be provided.

The grading of adverse events will be based on the guidelines provided in the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

#### 9.6.3 Laboratory Test Results

The subject listing of clinical laboratory will be provided for the full analysis set. The analyses of safety laboratory data for Troponin will be included as summary statistics over time by dose level



Protocol Number: 20200392

Date: 10 May 2024 

#### 9.6.4 Vital Signs

The listing of vital signs including systolic/diastolic blood pressure, heart rate, respiratory rate and temperature will be provided.

#### 9.6.5 Physical Measurements

The subject listing will be provided which will include parameters of physical measurements.

#### 9.6.6 Electrocardiogram

The listing of all on-study ECG data will be provided.

#### 9.6.7 Antibody Formation

No summary tables or listing will be provided.

#### 9.6.8 Exposure to Investigational Product

The subject listings will be provided with IP start and end date. The listing will also include planned dose, actual dose and reason for change or withheld of the planned dose.

### 9.6.9 Exposure to Non-investigational Product(s)/Auxiliary Medicinal Product(s)

NA

#### 9.6.10 Exposure to Concomitant Medication

No summary tables and listings will be provided.

#### 9.7 Other Analyses

#### 9.7.1.1.1 Pharmacokinetic Analyses

The analysis of pharmacokinetic endpoints will include data from all subjects who have received at least 1 dose of the investigational product and have at least 1 pharmacokinetic sample collected.

PK parameters for AMG 176 including, but not limited to, maximum observed concentration (Cmax), area under the concentration-time curve (AUC) and half-life (t1/2) will be estimated, if feasible.

## 9.7.2 Analyses of Pharmacokinetic or Pharmacokinetic/Pharmacodynamic Endpoints

NA

#### 9.7.3 Analyses of Clinical Outcome Assessments

NA



Protocol Number: 20200392

Date: 10 May 2024 

#### 9.7.4 Analyses of Health Economic Endpoints

NA

9.7.5

NA

#### 10. Changes From Protocol-specified Analyses

During the initial development of this document, it was realized that there are protocolspecified analyses that cannot be implemented/performed and the protocol is not required to be amended. Following changes are required-

- Though protocol states that the Uniform Response criteria were used for deriving the responses; however, International Working Group MDS Response Criteria (2006) (Appendix E) were used to classify responses for patients with MDS (based on NCCN guidelines Jan 2024). No patients with CMML were enrolled.
- Tables based on the primary analysis endpoints and secondary endpoints will not be generated due to the limited number of subjects and early close out of the study.
   These changes will also be documented in the Clinical Study Report.

Primary endpoints will not be analyzed using tables; however, listings will be provided only for clinical laboratory tests, vital signs, ECG, and adverse events including DLTs, treatment-related and treatment-emergent adverse events.

 Part 1A – QW Monotherapy (Dose Exploration)- Incidence of dose limiting toxicities (DLTs), treatment-related, treatment-emergent adverse events and clinically significant changes in vital signs, electrocardiogram (ECGs), and clinical laboratory tests.

No analysis will be performed for below secondary endpoints:

- Part 1B QW Combination Therapy (Dose Exploration) Overall response according to the IWG-MDS Response criteria for MDS/MPN (2006), EFS, time to response, and DOR
- 2. Part 2 QW Combination Therapy (Dose Expansion)
  - a. Time to transformation to Acute Myeloid Leukemia (AML)
  - b. Duration of Response (DOR)
  - c. Overall Survival (OS)
  - d. Time to Next MDS Treatment (TTNT)
  - e. EFS



Protocol Number: 20200392

Date: 10 May 2024 

#### 11. Literature Citations / References

Albitar M, Manshouri T, Shen Y, et al. Myelodysplastic syndrome is not merely "preleukemia". *Blood*. 2002;100(3):791-798.

AMG 176 Investigator's Brochure. Thousand Oaks, CA. Amgen Inc.

Ashkenazi A, Fairbrother WJ, Leverson JD, Souers AJ. From basic apoptosis discoveries to advanced selective BCL-2 family inhibitors. Nat Rev Drug Discov. 2017;16(4):273-284.

Bejar R, Steensma DP. Recent developments in myelodysplastic syndromes. *Blood*. 2014;124:2793-2803.

Beroukhim R, Mermel CH, Porter D, et al. "The landscape of somatic copy-number alteration across human cancers." *Nature*. 2010;463(7283):899-905.

Bose P, Grant S. MCL1 as a therapeutic target in acute myelogenous leukemia (AML). *Leukemia Research Reports*. 2013;2(1):12-14.

Caenepeel S, Brown SP, Belmontes B, et al. AMG 176, a selective MCL1 inhibitor, is effective in Hematological Cancer models alone and in combination with established therapies. *Cancer Discovery*. 2018;8:1582–1597.

Cairo MS, Bishop M. Tumour lysis syndrome: new therapeutic strategies and classification. *Br J Haematol.* 2004;127(1):3-11.

Cheson BD, Greenberg PL. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. *Blood.* 2006; 108 (2): 419-425.

Coiffier B, Altman A, Pui CH, et al. Guidelines for the management of pediatric and adult tumor lysis syndrome: an evidence-based review. *J Clin Oncol*. 2008;26(16):2767-2778.

Czabotar PE, Lessene G, Strasser A, Adams JM. Control of apoptosis by the BCL-2 protein family: implications for physiology and therapy. *Nat Rev Mol Cell Biol*. 2014;15(1):49-63.

Doll DC, List AF. Myelodysplastic syndromes. West J Med. 1989;151(2):161-167.

Fenaux P, Mufti GJ, Hellstrom-Lindberg E, et al. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. *Lancet Oncol*. 2009;10(3):223-232.

Fouad YA, Aanei C. Revisiting the hallmarks of cancer. *Am J Cancer Res.* 2017;7(5):1016-1036.

Glaser SP, Lee EF, Trounson E, et al. Anti-apoptotic Mcl-1 is essential for the development and sustained growth of acute myeloid leukemia. *Genes Dev.* 2012;26(2):120-125.

Greenberg P, Cox C, LeBeau MM, et al. International scoring system for evaluating prognosis in myelodysplastic syndromes. *Blood*. 1997;89(6):2079-2088.

Greenberg PL, Tuechler H, Schanz J, et al. Revised international prognostic scoring system for myelodysplastic syndromes. *Blood*. 2012;120(12):2454-2465.

Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000;100(1):57-70.



Protocol Number: 20200392

Date: 10 May 2024 

International Committee of Medical Journal Editors, Uniform Requirements for Manuscripts Submitted to Biomedical Journals: Writing and Editing for Biomedical Publication. 2013. http://www.icmje.org

International Conference on Harmonisation; S9 Guidance on Nonclinical Evaluation for Anticancer Pharmaceuticals. Fed Regist. 2010;Mar 8;75(44):10487-10488.

Jabbour E, Garcia-Manero G, Batty N, et al. Outcome of patients with myelodysplastic syndrome after failure of decitabine therapy. *Cancer*. 2010;116(16):3830-3834.

Ji Y, Liu P, Li Yisheng, Bekele BN. A modified toxicity probability interval method for dose-finding trials. *Clinical Trials*. 2010; 7:653-663.

Kadia TM, Jabbour E, Kantarjian H. Failure of hypomethylating agent-based therapy in myelodysplastic syndromes. *Semin Oncol.* 2011; 38(5):682-692.

Kantarjian H, Issa JP, Rosenfeld CS, et al. Decitabine improves patient outcomes in myelodysplastic syndromes: results of a phase III randomized study. *Cancer*. 2006;106(8):1794-1803.

Kasper S, Breitenbuecher F, Heidel F, et al. Targeting MCL1 sensitizes FLT3-ITD-positive leukemias to cytotoxic therapies. *Blood Cancer J.* 2012;2:e60.

Kaufmann SH, Karp JE, Svingen PA, et al. Elevated Expression of the Apoptotic Regulator MCL1 at the Time of Leukemic Relapse. *Blood*. 1998;91(3):991-1000.

Kotschy A, Szlavik Z, Murray J, et al. The MCL1 inhibitor S63845 is tolerable and effective in diverse cancer models. *Nature*. 2016;538(7626):477-482.

Kozopas KM, Yang T, Buchan HL, Zhou P, Craig RW. MCL1, a gene expressed in programmed myeloid cell differentiation, has sequence similarity to BCL2. *Proc Natl Acad Sci U S A*. 1993;90(8):3516-3520.

List AF. New agents in the treatment of MDS. *Clin Adv Hematol Oncol*. 2005;3(11):832-834.

Ma X, Does M, Raza A, Mayne ST. Myelodysplastic syndromes: incidence and survival in the United States. *Cancer*. 2007;109(8):1536-1542.

Merino D, Whittle JR, Vaillant F, et al. Synergistic action of the MCL-1 inhibitor S63845 with current therapies in preclinical models of triple-negative and HER2-amplified breast cancer. *Sci Transl Med*. 2017;9(401).

Mesa RA, personal communication, 2014.

Peperzak V, Vikström I, Walker J, et al. MCL1 is essential for the survival of plasma cells. *Nat Immunol*. 2013;14(3):290-297.

Prebet T, Gore SD, Esterni B, et al. Outcome of high-risk myelodysplastic syndrome after azacitidine treatment failure. *J Clin Oncol.* 2011;29(24):3322-3327.

Roberts AW, Davids MS, Pagel JM, et al. Targeting BCL2 with venetoclax in relapsed chronic lymphocytic leukemia. *N Engl J Med*. 2016;374:311-322. DOI: 10.1056/NEJMoa1513257.

Steensma DP. Can hypomethylating agents provide a platform for curative therapy in myelodysplastic syndromes? *Best Pract Res Clin Haematol*. 2012;25(4):443-451.

Strasser A, Cory S, Adams JM. Deciphering the rules of programmed cell death to improve therapy of cancer and other diseases. *EMBO J.* 2011;30(18):3667-3683.



Protocol Number: 20200392

Date: 10 May 2024 

Thall PF, Simon RM, Estey EH. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes. *Stat Med*. 1995;14(4):357-79.

Thomas RL, Roberts DJ, Kubli DA, et al. Loss of MCL-1 leads to impaired autophagy and rapid development of heart failure. *Genes Dev.* 2013;27(12):1365-1377.

van Delft MF, Wei AH, Mason KD, et al. The BH3 mimetic ABT-737 targets selective Bcl-2 proteins and efficiently induces apoptosis via Bak/Bax if Mcl-1 is neutralized. *Cancer Cell.* 2006;10(5):389-399.

Wang X, Bathina M, Lynch J, et al. Deletion of MCL-1 causes lethal cardiac failure and mitochondrial dysfunction. *Genes Dev.* 2013;27(12):1351-1364.

Wertz IE, Kusam S, Lam C, et al. Sensitivity to antitubulin chemotherapeutics is regulated by MCL1 and FBW7. *Nature*. 2011;471(7336):110-114

Xiang Z, Luo H, Payton J E, et al. Mcl1 haploinsufficiency protects mice from Myc-induced acute myeloid leukemia. *J Clin Investigation*. 2010;120(6):2109-2118.

Youle, RJ, Strasser A. The BCL2 protein family: opposing activities that mediate cell death. *Nat Rev Mol Cell Biol.* 2008;9(1):47-59

#### 12. Prioritization of Analyses

There is no prioritization of analyses.

#### 13. Data Not Covered by This Plan

The analyses of PK are not covered by this plan.



run;

Protocol Number: 20200392

Date: 10 May 2024 

#### 14. Appendices

#### **Appendix A. Code Fragments**

The ORR and its 95% CI can be calculated in SAS using PROC FREQ. The sample code is provided below, where RESP is the status of response (eg., 1=responder, 2=non-responder). The CI using the exact method can be found in the OUT data labeled as 'Exact Conf Limits'.

proc freq data=TEST; tables RESP / binomial alpha=0.05; ods output Binomial=OUT;



Protocol Number: 20200392

Date: 10 May 2024 

#### Appendix B. Modified Toxicity Probability Interval Design

A modified Toxicity Probability Interval (mTPI) design will be used to guide dose exploration. The OBD/MSBED is defined as the minimum safe and biologically effective combination dose with a probability of DLT lower than or close to a targeted toxicity probability of 0.2. The doses are considered close to the OBD if the toxicity probabilities belong to the proper dosing interval (0.25, 0.35) which corresponds to staying at the current dose (S). The underdosing interval is defined as (0, 0.25) in which the doses are deemed lower than the OBD and corresponds to a dose escalation (E). The overdosing interval is (0.35, 1) in which the doses are deemed higher than the OBD and corresponds to a dose de-escalation (D).

The dose-finding decisions are guided based on Bayesian decision rule by minimizing the posterior expected loss through calculating the Unit Probability Mass (UPM). At each dose level, the UPM is computed for the dosing intervals using the observed data enrolled at current dose. The dose-finding decision is determined as the interval with maximum UPM. A set of independent and non-informative prior Beta (1,1) is used for each dose level, which provides equal prior expected loss for the decisions (Ji et al, 2010). Dose escalation will not occur unless at least 6 subjects are treated at the current dose level. In addition, any dose whose posterior probability of toxicity is greater than the target toxicity exceeds 80% will be considered as unacceptable toxicity. This dose and higher doses will not be used again in the trial. Dose exploration will continue until either the maximum number of subjects (up to 30 subjects in monotherapy part and up to 30 subjects in combination therapy part) are treated or all doses are determined to be intolerable.



Protocol Number: 20200392

Date: 10 May 2024 

#### Appendix C. Last Known Alive Date

For subjects who do not have death date available i.e., subject was alive throughout, derive last known alive date as the latest of all the date variables below:

- 1. Events form: Date Started, Date Ended or Resulted in Death, hospitalization admission date, hospitalization date discharged.
- Date collected on Chemistry (Local lab), Chemistry (Local lab) (Unsched), Coagulation (Local Lab), Coagulation (Local Lab) (Unsched), Hematology (Local Lab), Hematology (Local Lab) (Unsched), Urinalysis (Local Lab), Urinalysis (Local Lab) (Unsched), Immunology (Local Lab), Reproductive Status and Pregnancy Test (Local Lab), Male Reproductive Status, Liver Biopsy Results, Liver Biopsy - Abnormal Findings, Liver Biopsy - Abnormal Architecture Findings, Liver Biopsy - Abnormal Liver Cell or Hepatocyte Findings, Liver Biopsy - Liver Cell or Hepatocyte Inclusion or Vacuole Types, Liver Biopsy - Hepatocyte or Liver Cell Nuclear Abnormality Types, Liver Biopsy - Liver or Lobular Infiltrate Types, Liver Biopsy - Portal Tract Inflammation Types, Liver Biopsy -Abnormal Bile Duct Findings, Liver Biopsy - Abnormal Portal Vein Findings, Liver Biopsy - Liver Infection Findings, Liver Biopsy - Parasite or Ova Findings, Liver Biopsy -Histological Staining or Additional Study Details, Liver Imaging Results, Hepatic Event Labs, Chemistry (Local Lab) (DILI), Coagulation (Local Lab) (DILI), Hematology (Local Lab) (DILI), Immunology (Local Lab) (DILI), Toxicology (Local Lab) (DILI), Chemistry (Local Lab) (Non-TP), Hematology (Local Lab) (Non-TP), Urinalysis (Local Lab) (Non-TP), Coagulation (Local Lab) (Non-TP),

(Non-TP) (Cardiac monitoring tests), Chemistry (Local Lab) (TLS monitoring tests), Chemistry (Local Lab) (Cardiac monitoring tests), Bone Marrow Aspirate for MDS, Chemistry (Local Lab) (Unsched) (TLS monitoring tests), Chemistry (Local Lab) (Unsched) (Cardiac monitoring tests), Hematology (Local Lab) (Peripheral Blood Counts), Hematology (Local Lab) (Unsched) (Peripheral Blood Counts), Hematology (Local Lab) (Peripheral Blood Counts) (Non-TP) forms.

- Date first taken, Date last taken on the Concomitant medications, Other Protocol Required Therapy (Allopurinol or equivalent), Anti-Cancer Therapies (On Study) forms.
- 4. Date performed on CT or MRI, ECOG performance status, Electrocardiogram Triplicate (On-study), Electrocardiogram (on-study), Procedure, Transfusions, NYHA Classification, Vital signs, Vital Signs (DILI), MUGA Scan or Echocardiogram, MUGA Scan or Echocardiogram (DILI), Electrocardiogram (On-study) (Non-TP),



Protocol Number: 20200392

Date: 10 May 2024 

Electrocardiogram - Triplicate (On-study) (Non-TP), Vital Signs Log (VS200), Vital Signs Log (VS200) (Non-TP) forms.

- 5. Date subject has ended IP, End of Investigational Product Administration, End of Non-Investigational Product Administration (Azacitidine), End of Safety Follow-up, EOS forms only if the status is not dead or lost to follow-up.
- 6. Hospitalization admission and dfischarge dates on hospitalization form
- 7. Date first taken, Date last taken, Progression Date, Best Response Date on the Anticancer therapies form.
- 8. Start and stop dates on Investigational Product administration, Non- Investigational Product Administration (Azacitidine) forms.
- 9. Date of examination on physical measurement, Physical Measurement (Weight), Physical Measurement (Height/Weight/BMI C) forms.
- 10. Date consent signed, Date consent withdrawn on additional consents/withdrawals of consent form
- 11. Date of contact/search, subject status date on the Survival Status form if the subject status is not unknown.
- 12. Date of assessment on Disease Response (MDS) form.
- 13. All the date fields on Best Overall Response/Progression form.
- 14. All dates from NDB data.



Protocol Number: 20200392

Date: 10 May 2024 

## Appendix D. Handling of Dates, Incomplete Dates and Missing Dates Imputation Rules for Partial or Missing Start Dates

The reference date for the following rules is the date of first dose of study drug.

| | | Stop Date | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Complete: | | Partial:<br>yyyymm | | Partial: | | Missing |
| Start Date | | < 1 <sup>st</sup><br>dose | ≥ 1 <sup>st</sup><br>dose | < 1 <sup>st</sup><br>dose<br>yyyymm | ≥ 1 <sup>st</sup><br>dose<br><i>yyyymm</i> | < 1 <sup>st</sup><br>dose<br><i>yyyy</i> | ≥ 1 <sup>st</sup><br>dose<br><i>yyyy</i> | |
| Partial: | = 1 <sup>st</sup> dose | 2 | 1 | n/a | 1 | n/a | 1 | 1 |
| уууутт | ≠ 1 <sup>st</sup> dose | 2 | 2 | 2 | 2 | 2 | 2 | 2 |
| Partial: | = 1 <sup>st</sup> dose | 3 | 1 | 3 | 1 | n/a | 1 | 1 |
| | ≠ 1 <sup>st</sup> dose | | 3 | | 3 | 3 | 3 | 3 |
| Missing | | 4 | 1 | 4 | 1 | 4 | 1 | 1 |

<sup>1=</sup>Impute the date of first dose; 2=Impute the first of the month; 3=Impute January 1 of the year; 4=Impute January 1 of the stop year

Note: For subjects who were never treated (first dose date is missing), partial start dates will be set to the first day of the partial month or first day of year if month is also missing.

#### Imputation Rules for Partial or Missing Stop Dates

Initial imputation

- If the month and year are present, impute the last day of that month.
- If only the year is present, impute December 31 of that year.
- If the stop date is entirely missing, assume the event or medication is ongoing.

If the imputed stop date is before the start date, set stop date to missing.

If the imputed stop date is after the death date, impute as death date.

#### Imputation Rules for Partial or Missing Death Dates

If death year and month are available but day is missing:

- If yyyymm for the date last known to be alive equals yyyymm for death date, set death date to the day after the date last known to be alive.
- If yyyymm for the date last known to be alive is less than the yyyymm for death date, set death date to the first day of the death month.



Protocol Number: 20200392

Date: 10 May 2024 

• If yyyymm for the date last known to be alive is greater than yyyymm for death date, assume date last known to be alive is in error, set death date to the first day of the death month.

If month and day are missing and year of death is known:

- If yyyy for the date last known to be alive equals yyyy for death date, set death date to the day after last known to be alive date.
- If yyyy for the date last known to be alive is less than yyyy for death date, set death date to the first day of the death year.
- If yyyy for the date last known to be alive is greater than yyyy for death date, assume
  date last known to be alive is in error, set death date to the first day of the death
  year.

If a death occurred and a death date is totally missing:

• Do not impute and censor the subject survival time.



Protocol Number: 20200392

Date: 10 May 2024 

# Appendix E. MDS Diagnostic and Response Criteria Proposed modified International Working Group response criteria for altering natural history of MDS

| Category | Response criteria (responses must last at least 4 wk) |
|---|---|
| Complete<br>remission | Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines* |
| | Persistent dysplasia will be noted*† |
| | Peripheral blood‡ |
| | Hgb ≥ 11 g/dL |
| | Platelets $\ge 100 \times 10^9 / L$ |
| | Neutrophils ≥ $1.0 \times 10^9/L^{\uparrow}$ |
| | Blasts 0% |
| Partial remission | All CR criteria if abnormal before treatment except: |
| | Bone marrow blasts decreased by $\geq 50\%$ over pretreatment but still > $5\%$ |
| | Cellularity and morphology not relevant |
| Marrow CR† | Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment |
| | Peripheral blood: if HI responses, they will be noted in addition to marrow CR† |
| Stable disease | Failure to achieve at least PR, but no evidence of progression for > 8 wks |
| Failure | Death during treatment or disease progression characterized by worsening of cytopenias, increase in percentage of bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment |
| Relapse after CR<br>or PR | At least 1 of the following: |
| | Return to pretreatment bone marrow blast percentage |
| | Decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets |
| | Reduction in Hgb concentration by $\geq 1.5$ g/dL or transfusion dependence |
| Cytogenetic | Complete |
| | Disappearance of the chromosomal abnormality without appearance of new ones |
| | Partial |
| | At least 50% reduction of the chromosomal abnormality |
| Disease<br>progression | For patients with: |
| | Less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts |
| 1<br>2<br>A | 5%-10% blasts: ≥ 50% increase to > 10% blasts |
| | 10%-20% blasts: ≥ 50% increase to > 20% blasts |
| | 20%-30% blasts: ≥ 50% increase to > 30% blasts |
| | Any of the following: |
| | At least 50% decrement from maximum remission/response in granulocytes or platelets |
| | Reduction in Hgb by $\geq 2$ g/dL |
| | Transfusion dependence |

